CLINICAL TRIAL: NCT05690126
Title: Investigation of the Effect of Saffron Extract Supplementation on Emotional Well-being Alterations in Healthy Volunteers: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Effect of Saffron Extract Supplementation on Emotional Well-being Alterations
Acronym: SAFFROMFOOD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022-A01556-37
Record Dates: First submitted 2022-12-21; First posted 2023-01-19 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Mood Disturbance
Keywords: Saffron extract; Depressive Symptoms; Fatigue; Emotional wellbeing; Sleep quality; Anxiety; Inflammation
MeSH Terms: conditions — Depression; Fatigue; Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Inflammation | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saffron extract (Active Comparator): Daily, two dietary supplements (Saffron extract) will be taken orally with water, the first one at breakfast and the second one at dinner.
  Dietary supplements in capsule form
  Interventions: Dietary Supplement: Saffron extract
- Placebo (Placebo Comparator): Daily, two dietary supplements (Maltodextrin) will be taken orally with water, the first one at breakfast and the second at dinner.
  Dietary supplements in capsule form
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Saffron extract — Food supplements are taken during 6 weeks by healthy volunteers
  Arms: Saffron extract
Dietary Supplement: Maltodextrin — Food supplements are taken during 6 weeks by healthy volunteers
  Arms: Placebo

SUMMARY:
This study aims to test whether a saffron extract represents a good candidate to improve emotional well-being in subjects with subclinical symptoms of depression, fatigue, stress or anxiety. Given that mild depression, both subclinical and chronic, was shown to predispose to major clinical depression, early initiation of neuroactive nutrient supplementation may be useful to prevent or counteract the onset of chronic depression.

The main objective of this study is to evaluate the efficacy of nutritional supplementation with saffron extract during 6 weeks in alleviating emotional well-being alterations in healthy adults presenting subclinical symptoms of depressed mood, anxiety, fatigue and/or stress.

The secondary objectives are to assess the impact of saffron extract supplementation on the mood and neurovegetative components of emotional well-being and quality of life, namely:

* depressive and anxious symptoms;
* neurovegetative symptoms (fatigue, sleep quality);
* perceived stress and quality of life.

The exploratory objectives correspond to the biological assays for the evaluation of

* the stress response system (stress hormones);
* the inflammatory status;
* saffron metabolites;
* metabolome.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (as determines by medical history and clinical examination);
* Male or female between 18 and 50 years of age;
* Body Mass Index (BMI) 18.5 ≤ BMI < 30 kg/ m2;
* Subject with subclinical symptoms of depressed mood, anxiety, fatigue and/or stress, as determined by the presence of at least 6 or more symptoms of moderate intensity among the 18 symptoms listed in the modified neurotoxicity scale (NRS).
* Subject able and willing to participate to the study by complying with the protocol procedures as confirmed by his dated and signed informed consent form;
* Person affiliated or benefiting from a social security scheme.

Exclusion Criteria:

* Psychiatric comorbidity determined with the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM5) or history of psychiatric illness;
* Neurodegenerative pathology (Alzheimer's disease, Parkinson's disease, dementia);
* Cardio-metabolic diseases (cardiovascular diseases, type 1 or 2 diabetes...);
* Untreated or unstabilised hypertension;
* Severe chronic diseases (cancer, severe chronic pain, HIV, hepatitis, kidney disease, autoimmune diseases, etc.);
* Chronic inflammatory diseases (Crohn's disease, coeliac disease, rheumatoid arthritis, etc.);
* Pathologies likely to act on the Hypothalamus-Pituitary-Adrenal (HPA) axis or the adrenal cortical metabolism (e.g.: Cushing syndrome);
* Untreated and/or unstabilised thyroid diseases (hypo/hyperthyroidism, Graves' disease...);
* Subjects treated during the previous 6 months or being currently treated with psychotropic drugs prescribed and/or recommended for anxiety, depression, sleep disorders and generally for any neurological or psychological type of manifestation.

The same applies to:

* Drugs likely to have direct or indirect effects on psychiatric symptoms, notably regular use of corticoids or steroidal anti-inflammatories (e.g. Betamethasone, Cortivazol, Dexamethasone, Methylprednisolone, Prednisolone, Prednisone, Tetracosactide, Triamcinolone, etc.);
* Any drug treatment aimed at improving or maintaining cognitive functions (e.g. Aricept, Exelon, Reminyl, Ebixa etc.);
* Food supplements during the last 3 months prior to participation in this study.
* Personal or professional event with potential severe impact on the subject's emotional and/or psychological state within the last 8 weeks (e.g. but not limited to: change of job function/position, death of a family member, divorce, surgery, accident, etc.);
* Use of antibiotic treatment (<2 months);
* Recent treatment with non-steroidal anti-inflammatory drugs (<1 month);
* Bariatric surgery;
* Subject with asthma, allergies (allergic rhinitis, atopic dermatitis);
* Any documented or suspected food allergy to any component of the study products.
* Drug dependence (except tobacco);
* Tobacco use of more than 20 cigarettes per day;
* Consumption of large quantities of coffee, tea, chocolate (more than 5 cups of coffee or tea and more than 20 g of dark chocolate per day) or regular daily consumption of herbal infusions with relaxing or hypnotic properties [e.g. chamomile, valerian, passionflower etc];
* Alcohol abuse (maximum 2 drinks per day, maximum 10 drinks per week with several days of abstinence) or recreational drug use based on the participant's declaration;
* Eating disorders: anorexia and bulimia or unstable diet;
* Xerostomia or other conditions that may make saliva collection impossible;
* Subjects working shifts or in extreme conditions (e.g. cold storage);
* Intense physical activity: more than 10 hours per week of intense physical activity, or significant change in physical activity within the last 2 months, or physical activity likely to be modified within the next 6 weeks. Examples of moderate to vigorous physical activity are: carrying heavy loads, playing tennis (singles or doubles), combat sports, "fast" swimming, jogging etc. Walking is not considered a moderate intensity physical activity.
* Subjects whose language skills do not allow them to understand the questionnaires;
* Disability (psychological, visual, psychomotor, linguistic...) likely to compromise to understand and sign the consent form and to complete self-questionnaires during the study.
* Subject participating in another interventional study or being in the exclusion period of a previous clinical trial;
* Subject receiving more than 4500 euros as indemnities for participation in biomedical research within the 12 last months, including indemnities for the present study;
* Women who are pregnant, intend to become pregnant during the study or are breastfeeding.
* Hormonal state that may induce a fluctuating emotional state during the study, such as, postpartum (< 6 months after delivery) and peri-menopause (irregular menstrual cycle, hot flashes, feeling of swelling, breast tension).
* Subjects under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in emotional well-being composite score | Baseline (V1) and 6 weeks (V2)
  The primary endpoint is the change from baseline (V1) to 6 weeks (V2) in the composite Z-score of emotional well-being combining three components: depression (BDI score), anxiety (STAI state score) and fatigue (MFI score).

SECONDARY OUTCOMES:
Change in mood | Baseline (V1) and 6 weeks (V2)
  Beck Depression Inventory (score 0-39).
Change in anxiety | Baseline (V1) and 6 weeks (V2)
  State-Trait Anxiety Inventory (score 20-80).
Change in stress | Baseline (V1) and 6 weeks (V2)
  Visual analog scale for stress (score 0 to 10).
Change in fatigue | Baseline (V1) and 6 weeks (V2)
  Multidimensional Fatigue Inventory (MFI) (score 20-100).
Change in sleep quality | Baseline (V1) and 6 weeks (V2)
  The Pittsburgh Sleep Quality Index (PSQI) (score 0 to 21).
Change in neurovegetative symptomatology | Baseline (V1) and 6 weeks (V2)
  Neurotoxic rating scale (NRS) (score 0 to 152).
Change in quality of life | Baseline (V1) and 6 weeks (V2)
  Medical Outcome Study Short Form 12 (SF-12) (score 0 to 100).
Change in dietary intake | Baseline (V1) and 6 weeks (V2)
  Subjects will complete a food diary in which they will register all the food and drinks consumed during 3 defined days (two weekdays and one weekend day).
  The Programme national nutrition santé (PNNS) questionnaire is a non-quantitative food frequency questionnaire. The 12 items are based on the recommendations of the French National Nutrition and Health.
Change in stress response system | Baseline (V1) and 6 weeks (V2)
  Salivary cortisol as a measure of the stress response system.
Change in inflammatory markers | Baseline (V1) and 6 weeks (V2)
  Blood levels of acute phase proteins and cytokines.
Change in oxidative stress | Baseline (V1) and 6 weeks (V2)
  Blood oxidative stress markers such as malondialdehyde (MDA), total antioxidant capacity (TCA) and superoxide dismutase (SOD) levels.
Change in saffron metabolites | Baseline (V1) and 6 weeks (V2)
  Blood and urine polyphenols and carotenoids levels.
Change in metabolome | Baseline (V1) and 6 weeks (V2)
  Untargeted metabolomics analysis in blood and urine samples using nuclear magnetic resonance (NMR) and/or liquid chromatography-mass spectrometry (LC-MS).
Change in lipid profile | Baseline (V1) and 6 weeks (V2)
  Lipids profile in red blood cells.

CONTACTS AND LOCATIONS:
Overall Officials: Lucile Capuron, PhD, Study Director — INRAE-Laboratory of Nutrition And Integrative Neurobiology (NutriNeuro Lab)
Locations (1):
- CEN Experimental, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amadieu C, Leyrolle Q, Farneti M, Anesi A, Bruchet E, Montet J, Dexpert S, Gaudout D, Mattivi F, Pourtau L, Castanon N, Capuron L. Effect of saffron extract supplementation on mood in healthy adults with subclinical symptoms of depression: a randomized, double-blind placebo-controlled study. Am J Clin Nutr. 2025 Dec;122(6):1625-1635. doi: 10.1016/j.ajcnut.2025.09.050. Epub 2025 Oct 3. PMID 41047129